CLINICAL TRIAL: NCT06588036
Title: A Comprehensive Analysis of the Comparative Efficacy of Multimodal Diarrhea Therapies
Brief Title: A Comprehensive Analysis of the Comparative Efficacy of Multimodal Diarrhea Therapies in the Paediatric Population
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Multan (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Aamir Aslam Awan, Assistant Professor, Combined Military Hospital Multan
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CMHMultan
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: To Assess the Mean Time of Resolution of Diarrhea
MeSH Terms: interventions — Prebiotics; Zinc; Time; smecta

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): : Group 1 receiving zinc and probiotic supplementation, Group 2 receiving zinc, probiotic, and prebiotics. Group 3 receiving zinc, probiotics, and anti-secretory agents, and Group 4 receiving zinc, probiotic, anti-secretory agents, and adsorbents.
  Interventions: Drug: Prebiotic; Other: Duration
- Duration of diarrhea (Active Comparator): This will showcase the duration of diarrhea that the pediatric population had before receiving treatment.
  Interventions: Drug: Prebiotic; Drug: Smecta

INTERVENTIONS:
Drug: Prebiotic — . The primary outcome measure will be the mean time from the initiation of treatment to the resolution of diarrhea symptoms. This objective seeks to provide evidence-based insights into the optimal management strategies for childhood diarrhea and inform clinical practice guidelines.
  Other Names: zinc; adsorbent; anti-secretory
Other: Duration — every participant is alloted a group based on RCT.
  Arms: Intervention Group
Drug: Smecta — Group 4 will be given smecta scahet
  Arms: Duration of diarrhea

SUMMARY:
The objective of this research is to assess the mean time of resolution of diarrhea in pediatric patients receiving different intervention combinations for the management of acute diarrhea. Specifically, the study aims to compare the effectiveness of four intervention groups: Group 1 receiving zinc and probiotic supplementation, Group 2 receiving zinc, probiotic, and prebiotics. Group 3 receiving zinc, probiotics, and anti-secretory agents, and Group 4 receiving zinc, probiotic, anti-secretory agents, and adsorbents. The primary outcome measure will be the mean time from the initiation of treatment to the resolution of diarrhea symptoms. This objective seeks to provide evidence-based insights into the optimal management strategies for childhood diarrhea and inform clinical practice guidelines.

DETAILED DESCRIPTION:
This study will employ a randomized controlled trial (RCT) design and will be conducted at the Combined Military Hospital (CMH) in Multan, Pakistan, from September 15, 2024, to December 15, 2024. A total of 100 patients will be included, with approximately 25 patients allocated to each intervention group. The sampling technique will be convenience sampling, where patients meeting the inclusion criteria and presenting during the study period will be recruited.

The main study variables include the intervention groups-Group 1: zinc and probiotic, Group 2: zinc, probiotic, and prebiotics, Group 3: zinc, probiotics, and anti-secretory, and Group 4: zinc, probiotic, anti-secretory, and adsorbent-time to resolution of diarrhea, and clinical outcomes. Data will be collected through caregiver interviews, clinical examinations, and a review of medical records. A structured questionnaire or proforma will be used to gather relevant information from patients and caregivers regarding demographic characteristics, clinical presentation, interventions received, and outcomes.

**Data Analysis Procedure:** Statistical analysis will be conducted using SPSS software, version 28.0 (IBM Corp., Armonk, NY). Both quantitative and qualitative data will be analyzed, with descriptive statistics such as mean, median, standard deviation, and frequency distributions used to summarize the demographic and clinical characteristics of the study population. For comparing outcomes between intervention groups, inferential statistical tests such as ANOVA for continuous variables and the Chi-square test for categorical variables will be employed, depending on the nature of the data. Confounding variables will be controlled through multivariate analysis, and a p-value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

* Pediatric patients, both male and female, aged 6 months to 5 years presenting with acute diarrhea at CMH Multan.
* Patients or caregivers willing to provide informed consent for participation in the study.

Exclusion Criteria:

* Pediatric Patients with chronic diarrhea or underlying gastrointestinal disorders.
* Pediatric Patients with severe dehydration requiring immediate medical intervention.
* Pediatric Patients with a history of allergy or intolerance to any of the study interventions.
* Pediatric Patients with severe comorbidities or immunocompromised status.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
resolution of diarrhea | 3 months
  mean time of resolution of diarrhea in different intervention groups

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad F Shafiq, Study Chair — CMH Multan

IPD SHARING:
Plan to Share IPD: No